CLINICAL TRIAL: NCT05039450
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study of Efruxifermin in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH) (Symmetry)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0103
Record Dates: First submitted 2021-07-29; First posted 2021-09-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- EFX 28 mg (Main Study) (Experimental)
  Interventions: Drug: EFX
- EFX 50 mg (Main Study) (Experimental)
  Interventions: Drug: EFX
- Placebo (Main Study) (Placebo Comparator)
  Interventions: Drug: Placebo
- EFX 50 mg (Cohort D) (Experimental)
  Interventions: Drug: EFX
- Placebo (Cohort D) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EFX — Investigational drug, Efruxifermin
  Arms: EFX 28 mg (Main Study); EFX 50 mg (Cohort D); EFX 50 mg (Main Study)
Drug: Placebo — Placebo
  Arms: Placebo (Cohort D); Placebo (Main Study)

SUMMARY:
This is a multi-center evaluation of efruxifermin (EFX) in a randomized, double-blind, placebo-controlled study in cirrhotic subjects with biopsy-proven F4 compensated NASH.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females between 18-75 years of age inclusive, based on the date of signing informed consent.
* Main Study Only: Previous history or presence of Type 2 diabetes or 2 out of 4 components of metabolic syndrome (obesity, dyslipidemia, elevated blood pressure, elevated fasting glucose).
* Main Study Only: Biopsy-proven compensated cirrhosis due to NASH.
* Cohort D Only: Diagnosis of type 2 diabetes
* Cohort D Only: Use of GLP-1R agonist for at least 90 days
* Cohort D Only: Biopsy-proven liver fibrosis stages 1, 2, or 3

Exclusion Criteria:

* Main Study Only: Weight loss > 10% in the 90 days prior to screening until randomization or from the time of collection of the liver biopsy used to assess subject eligibility until randomization, whichever is longer.
* Type 1 diabetes or uncontrolled Type 2 diabetes
* Cohort D Only: Weight loss > 5% in the 90 days prior to screening
* Cohort D Only: Presence of cirrhosis on liver biopsy

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Main: Change from baseline in fibrosis with no worsening steatohepatitis assessed by NASH CRN system | Week 36
  Proportion of subjects who achieve ≥ 1 stage improvement in fibrosis (based on NASH CRN fibrosis score) and no worsening of steatohepatitis at Week 36.

SECONDARY OUTCOMES:
Main: Resolution of NASH assessed by the NASH CRN system | Week 36, Week 96
  Proportion of subjects who achieve NASH resolution (defined as a NAS of 0-1 for inflammation and 0 for ballooning) as determined by the NASH CRN criteria at Week 36 and Week 96
Main: Fibrosis improvement with no worsening of NASH assessed by the NASH CRN system | Week 36, Week 96
  Proportion of subjects who achieve NASH resolution (defined as a NAS of 0-1 for inflammation and 0 for ballooning) and ≥ 1 stage improvement in fibrosis (based on NASH CRN fibrosis score) at Week 36 and Week 96
Main: Change from baseline in fibrosis in subjects with no worsening of steatohepatitis assessed by the NASH CRN system | Week 96
  Proportion of subjects who achieve ≥ 1 stage improvement in fibrosis (based on NASH CRN fibrosis score) and no worsening of steatohepatitis at Week 96
Main: Change from baseline in fibrosis in subjects with no worsening of steatohepatitis assessed by the NASH CRN system | Week 36, Week 96
  Proportion of subjects who achieve ≥ 1 stage improvement in fibrosis (based on NASH CRN fibrosis score) at Week 36 and Week 96
Main: Change from baseline in non-invasive markers of fibrosis | Week 36, Week 48, Week 72, Week 96
  Change from baseline in ELF score, Pro-C3 (ug/L),and liver stiffness assessed by liver elastography (kPa, CAP)
Main: Change from baseline in lipoproteins | Week 36, Week 48, Week 72, Week 96
  Change from baseline in Triglycerides (mg/dL), total cholesterol (mg/dL), HDL-C (mg/dL), non-HDL-C (mg/dL), and LDL-C (mg/dL)
Main: Change from baseline of markers in insulin sensitivity and glycemic control | Week 36, Week 48, Week 72, Week 96
  Change from baseline in HbA1c (%), C-peptide (ug/L), adiponectin (mg/L), insulin (mIU/L), and HOMA-IR
Main: Change from baseline in body weight | Week 36, Week 48, Week 96
  Change from baseline in body weight (kg)
Main: To assess the immunogenicity of EFX | Through Week 96
  Detect and measure ADA, including NAb, against EFX
Main: To assess the safety and tolerability of EFX | Through Week 96
  Safety and tolerability will be assessed through the reporting of AEs, clinical laboratory tests, ECGs, ultrasounds, vital sign assessments, and concomitant medication usage
Cohort D: To assess the safety and tolerability of EFX compared to placebo when added to an existing GLP-1R agonist in subjects with type 2 diabetes and liver fibrosis due to NASH | Through Week 12
  Safety and tolerability will be assessed through the reporting of AEs, clinical laboratory assessments, ECGs, ultrasounds, vital sign assessments, and concomitant medication usage

CONTACTS AND LOCATIONS:
Locations (44):
- United States (41):
  - Akero Clinical Study Site, Chandler, Arizona
  - Akero Clinical Study Site, Glendale, Arizona
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, North Little Rock, Arkansas
  - Akero Clinical Study Site, Fresno, California
  - Akero Clinical Study Site, Long Beach, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Pasadena, California
  - Akero Clinical Study Site, Englewood, Colorado
  - Akero Clinical Study Site, Clearwater, Florida
  - Akero Clinical Study Site, Fort Myers, Florida
  - Akero Clinical Study Site, Hialeah Gardens, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Miami Lakes, Florida
  - Akero Clinical Study Site, Ocala, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, South Bend, Indiana
  - Akero Clinical Study Site, Topeka, Kansas
  - Akero Clinical Study Site, Bastrop, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Las Vegas, Nevada
  - Akero Clinical Study Site, Concord, North Carolina
  - Akero Clinical Study Site, Fayetteville, North Carolina
  - Akero Clinical Study Site, Morehead City, North Carolina
  - Akero Clinical Study Site, Springboro, Ohio
  - Akero Clinical Study Site, Westlake, Ohio
  - Akero Clinical Study Site, Greenville, South Carolina
  - Akero Clinical Study Site, Greenwood, South Carolina
  - Akero Clinical Study Site, Summerville, South Carolina
  - Akero Clinical Study Site, Nashville, Tennessee
  - Akero Clinical Study Site, Austin, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, Houston, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, Waco, Texas
  - Akero Clinical Study Site, Webster, Texas
  - Akero Clinical Study Site, Wichita Falls, Texas
  - Akero Clinical Study Site, Ogden, Utah
  - Akero Clinical Study Site, Richmond, Virginia
- Mexico (2):
  - Akero Clinical Study Site, Mexico City
  - Akero Clinical Study Site, Monterrey
- Akero Clinical Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureddin M, Rinella ME, Chalasani NP, Neff GW, Lucas KJ, Rodriguez ME, Rudraraju M, Patil R, Behling C, Burch M, Chan DC, Tillman EJ, Zari A, de Temple B, Shringarpure R, Jain M, Rolph T, Cheng A, Yale K. Efruxifermin in Compensated Liver Cirrhosis Caused by MASH. N Engl J Med. 2025 Jun 26;392(24):2413-2424. doi: 10.1056/NEJMoa2502242. Epub 2025 May 9. PMID 40341827
- [Derived] Harrison SA, Frias JP, Lucas KJ, Reiss G, Neff G, Bollepalli S, Su Y, Chan D, Tillman EJ, Moulton A, de Temple B, Zari A, Shringarpure R, Rolph T, Cheng A, Yale K. Safety and Efficacy of Efruxifermin in Combination With a GLP-1 Receptor Agonist in Patients With NASH/MASH and Type 2 Diabetes in a Randomized Phase 2 Study. Clin Gastroenterol Hepatol. 2025 Jan;23(1):103-113. doi: 10.1016/j.cgh.2024.02.022. Epub 2024 Mar 4. PMID 38447814